CLINICAL TRIAL: NCT03591939
Title: Role of T-regulatory Cells in Type Two Diabetic Nephropathy
Brief Title: T-regulatory Cells in Diabetic Type Two Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, HSGalal, principal investigator, Assiut University
Other Study IDs: TRD
Record Dates: First submitted 2018-07-08; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Diabetic Nephropathy Type 2
MeSH Terms: interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: cases of Diabetic type two nephropathy
  Interventions: Diagnostic Test: laboratory test
- 2: controls of normal subjects
  Interventions: Diagnostic Test: laboratory test

INTERVENTIONS:
Diagnostic Test: laboratory test — role of T- regulatory cells in the patients of diabetic nephropathy

SUMMARY:
Diabetes mellitus is one of the most prevalent health problems worldwide. Diabetic nephropathy has become the leading cause of end-stage kidney disease worldwide and is associated with an increased cardiovascular risk.

Traditionally, metabolic and hemodynamic factors are the main causes of renal lesions in patients with type two diabetes mellitus and diabetic nephropathy , both considered non-immune diseases. Serial researches has demonstrated that diabetic nephropathy is a metabolic and hemodynamic disorder, with inflammation playing a vital role in the process.

DETAILED DESCRIPTION:
It has been reported that glomerular basement membranes from diabetic rats induced significantly greater amounts of Tumor necrotic factor-alpha and Interleukin-1 than when these cells were incubated with basement membranes from non-diabetic rats.

These new findings were the first to suggest that inflammatory cytokines may participate in the pathogenesis of diabetic nephropathy .Cluster of differentiation 4 cells are believed to play central roles in modulating immune responses. Tumor necrotic factor-alpha and Interleukin-6, and induce inflammation in the pathogenesis of autoimmune diseases.

T- regulatory cells exert immunosuppressive effects which are important on the maintenance of immune homeostasis by producing anti-inflammatory cytokines, such as Interleukin-10 and transforming growth factor-b.

Aim of this work is to the role of T regulatory cells :( Cluster of differentiation 4, Cluster of differentiation 25,Cluster of differentiation 127 , forkhead box P3 cells) in the different stages of diabetic nephropathy before hemodialysis initiation.

ELIGIBILITY:
Inclusion Criteria:

Adult patients above 20 years diagnosed with type 2 diabetes mellitus and have microalbuminuria, macroalbuminuria or renal impairment

Exclusion Criteria:

Patients with ischemic heart disease, any other autoimmune diseases, and Hepatitis C or B positive patients.

b-Patients with diabetic nephropathy on dialysis therapy c- Patients with any other causes for renal diseases such as glomerulonephritis

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects will be collected in a questionnaire form; from outpatient clinic in Assiut University hospital .These will be included in a file sheet for each subject : Age, Sex, Body height, weight and body mass index,Special habits ,fundus examination and neurological examination ,Blood pressure, pulse ,General and systematic examination Investigations will include; urine analysis, blood urea and serum creatinine, complete blood count, Fasting and 2 h post pranidal glucose levels
Sampling Method: Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
rate of patients with positive T-regulatory cells in blood | one week
  number of patients with diabetic type two nephropathy with positive T-regulatory cells in blood

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolf G. New insights into the pathophysiology of diabetic nephropathy: from haemodynamics to molecular pathology. Eur J Clin Invest. 2004 Dec;34(12):785-96. doi: 10.1111/j.1365-2362.2004.01429.x. PMID 15606719
- [Background] Rivero A, Mora C, Muros M, Garcia J, Herrera H, Navarro-Gonzalez JF. Pathogenic perspectives for the role of inflammation in diabetic nephropathy. Clin Sci (Lond). 2009 Mar;116(6):479-92. doi: 10.1042/CS20080394. PMID 19200057
- [Background] Hasegawa G, Nakano K, Sawada M, Uno K, Shibayama Y, Ienaga K, Kondo M. Possible role of tumor necrosis factor and interleukin-1 in the development of diabetic nephropathy. Kidney Int. 1991 Dec;40(6):1007-12. doi: 10.1038/ki.1991.308. PMID 1762301
- [Background] Adkins B, Leclerc C, Marshall-Clarke S. Neonatal adaptive immunity comes of age. Nat Rev Immunol. 2004 Jul;4(7):553-64. doi: 10.1038/nri1394. No abstract available. PMID 15229474
- [Background] Cheng X, Yu X, Ding YJ, Fu QQ, Xie JJ, Tang TT, Yao R, Chen Y, Liao YH. The Th17/Treg imbalance in patients with acute coronary syndrome. Clin Immunol. 2008 Apr;127(1):89-97. doi: 10.1016/j.clim.2008.01.009. Epub 2008 Feb 21. PMID 18294918
- [Background] Sakaguchi S, Ono M, Setoguchi R, Yagi H, Hori S, Fehervari Z, Shimizu J, Takahashi T, Nomura T. Foxp3+ CD25+ CD4+ natural regulatory T cells in dominant self-tolerance and autoimmune disease. Immunol Rev. 2006 Aug;212:8-27. doi: 10.1111/j.0105-2896.2006.00427.x. PMID 16903903